CLINICAL TRIAL: NCT05012202
Title: Validating a New Point-of-care Device for Estimation of Blood Count in Pregnant Women
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 21-0123
Record Dates: First submitted 2021-07-20; First posted 2021-08-19 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Blood Loss
Keywords: Vaginal delivery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Hemi device — A sample of vaginal blood will be collected following delivery and analyzed by the device to provide a hematocrit level, which will be masked to the clinical team.

SUMMARY:
Postpartum hemorrhage is a well-known complication of delivery and the leading cause of maternal mortality worldwide. In developed nations, a complete blood count (CBC) is commonly collected as a means to assess or base treatment for blood loss. The Hemi device is a point-of-care device designed to provide hematocrit, followed by the stage of hemorrhagic shock using artificial intelligence algorithms. The ultimate goal of the product is to provide an accurate hematocrit from easily attainable samples such as vaginal blood during hemorrhage to remove yet another barrier to access for actively bleeding women. The purpose of this study is to compare the hematocrit of vaginal blood using the Hemi device with standard venipuncture.

DETAILED DESCRIPTION:
This will be a prospective cohort study. The investigators will recruit 41 pregnant women admitted for delivery. Following delivery, a sample of vaginal blood will be collected and the Hemi device will be used to obtain hematocrit. These results will be masked to the clinical team until the time of data collection. A CBC will also be collected via venipuncture at this time. This study will be comparing hematocrit levels by standard clinical laboratory versus results from the device.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-50
* Admission for vaginal delivery
* Singleton pregnancy
* Term gestation (>=37 weeks)

Exclusion Criteria:

* Pregnant women < 18 years or > 50 years
* Incarcerated patients
* Patient unwilling or unable to provide consent
* Enrolled in another trial that may affect outcome

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes pregnant women admitted to the Labor & Delivery unit for delivery.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Hematocrit | During delivery
  Comparison of hematocrit from vaginal blood sample versus systemic sample

SECONDARY OUTCOMES:
Time to obtain results | During delivery
  Time to obtain hematocrit level results

CONTACTS AND LOCATIONS:
Locations (1):
- UTMB, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided